CLINICAL TRIAL: NCT06993324
Title: Awareness of Family With Down Syndrome Children About the Role of Physical Therapy Amongst Egyptian People
Brief Title: Awareness of Families With Down Syndrome Children About the Role of Physical Therapy in Egypt
Acronym: DS-AWARENESS
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Alaa Elsayed Atia Hassan Elkalla, Student Researcher, Cairo University
Other Study IDs: P.T.REC/012/005779
Record Dates: First submitted 2025-05-18; First posted 2025-05-28 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-08

CONDITIONS: Down Syndrome (DS)
Keywords: Awareness; Genetic Disorders; Physical Therapy; Egypt; Down Syndrome
MeSH Terms: conditions — Down Syndrome; Genetic Diseases, Inborn

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Families of Children with Down Syndrome: This group consists of family members (parents or primary caregivers) of children diagnosed with Down Syndrome. Participants will be surveyed to assess their awareness and knowledge about the role of physical therapy in managing developmental challenges associated with Down Syndrome. No interventions will be conducted as part of this study.

SUMMARY:
This study explores how much families with children who have Down Syndrome in Egypt know about the benefits and role of physical therapy. By understanding their awareness, hope to improve education and support so that these families can better access physical therapy services that can help improve their children's quality of life.

DETAILED DESCRIPTION:
This cross-sectional study aims to assess the awareness of families with children who have Down Syndrome regarding the role of physical therapy in Egypt. Data will be collected via a validated questionnaire distributed to family members to evaluate their knowledge and perceptions about physical therapy interventions. The study seeks to identify gaps in awareness and inform strategies for improving educational outreach and support for these families.

ELIGIBILITY:
Inclusion Criteria:

* Parents/guardians of children diagnosed with DS.
* Egyptian residents.
* Consent to participate in the study
* Aged 18 years or older

Exclusion Criteria:

* Families with children who have conditions other than DS.
* Participants who do not provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study includes family members and primary caregivers of children with Down Syndrome in Egypt. The participants will complete a questionnaire designed to assess their awareness of the role of physical therapy in managing developmental challenges.
Sampling Method: Non-Probability Sample
Enrollment: 240 (Actual)
Dates: Start 2025-04-05 (Actual); Primary Completion 2025-08-25 (Actual); Study Completion 2025-08-25 (Actual)

PRIMARY OUTCOMES:
Awareness Level of Families About the Role of Physical Therapy | "Baseline (single assessment using questionnaire at the beginning of the study)"
  This measure assesses the level of knowledge and awareness that family members of children with Down Syndrome have regarding physical therapy's benefits and role in improving their children's development and quality of life. It is evaluated through a validated questionnaire designed to capture understanding of physical therapy interventions and perceptions.

SECONDARY OUTCOMES:
Factors Influencing Awareness of Physical Therapy Among Families | "Baseline (single assessment using questionnaire at the beginning of the study)"
  This measure evaluates demographic, social, and educational factors that may affect the awareness levels of families with children who have Down Syndrome about physical therapy. It includes analysis of variables such as caregiver education level, access to healthcare information, and previous exposure to physical therapy services.

CONTACTS AND LOCATIONS:
Overall Officials: Maya G Aly, Assistant Professor, Study Director — Cairo University
Locations (1):
- Faculty of Physical Therapy, Cairo University, Giza, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared with other researchers to protect participant confidentiality and privacy. The data collected will only be used for the purpose of this study.